CLINICAL TRIAL: NCT02588937
Title: Active Drug Comparative Trial to Evaluate the Antiviral Activity and Safety in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 361HBV15017
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Entecavir, EntecaBell ODT., Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir

ARMS (2):
- EntecaBell ODT. (Experimental)
  Interventions: Drug: EntecaBell ODT. 0.5mg
- Baraclude Tab. (Active Comparator)
  Interventions: Drug: Baraclude Tab. 0.5mg

INTERVENTIONS:
Drug: EntecaBell ODT. 0.5mg
  Arms: EntecaBell ODT.
Drug: Baraclude Tab. 0.5mg
  Arms: Baraclude Tab.

SUMMARY:
The purpose of this study is to evaluate the antiviral activity and safety of EntecaBell ODT. in chronic hepatitis B Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 20 years old
2. Patients with Chronic Hepatitis B diagnosed
3. Patients who show positive HBsAg
4. Patients who show positive HBeAg or negative HBeAg
5. Patients who showed HBV DNA undetected(less than 300 copies/mL)
6. Patients who have administered Baraclude Tab. 0.5mg for 1~4 years
7. Patients who showed ALT less than 5 times of the upper limit in the normal range
8. Patient who decided to participate and signed on an informed consent form willingly

Exclusion Criteria:

1. Patients who have hepatitis C (HCV), hepatitis D (HDV), or human immunodeficiency virus (HIV)
2. Patients with a uncompensated liver disease who have at least one of the following values or signs

   * Total bilirubin > 2.5mg/dl
   * Prothrombin time delayed more than three seconds of upper limit in the normal range
   * Serum Albumin < 3 g/dL
   * A medical history of ascites, jaundice, hemorrhage by varix, hepatic encephalopathy, or other signs of liver function loss
3. Patients who are estimated to have hepatocellular carcinoma (HCC) through imaging examination or showed alpha-fetoprotein(AFP) more than 100 ng/mL
4. Patients who showed Creatinine Clearance < 50 mL/min by calculating Cockcroft-Gault equation
5. Patients who were not administered any anti-viral agents except Baraclude Tab.(Entecavir)
6. Administration of other Investigational Product within 30 days
7. History of malignant tumor within 5 years (including leukemia and lymphoma)
8. Patients who have a severe disease, such as heart failure, renal failure, and pancreatitis, decided by an investigator to have an effect on this clinical trial
9. Patients who have other hepatic diseases except hepatitis B
10. Administration immunosuppressants or corticosteroids over 2 weeks within 24 weeks
11. Patients who have to administer immunosuppressants or Nephrotoxic drugs, Hepatotoxic drugs for period of Clinical Trial
12. Pregnant, breast-feeding and childbearing age who don't use adequate contraception
13. Patients who are possible to decline daily function due to a mental disease or patients who are not able to understand the purpose and methods of this clinical trial
14. Patients who received an organ transplant or are going to received an organ transplant
15. Severe hypersensitivity to Entecavir
16. Another clinical condition in investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 300copies/mL) | 48 week

SECONDARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 300copies/mL) | 24 week
The Difference between the baseline and at the 24, 48 week of HBV DNA level(log10) | 24, 48 week
The rate of subjects who showed HBeAg serum loss | 24, 48 week
The rate of subjects who showed HBeAg seroconversion | 24, 48 week
The rate of subjects who showed HBsAg serum loss | 48 week
The rate of subjects who showed HBsAg seroconversion | 48 week
The rate of subjects who showed Virologic breakthrough | 12, 24, 48 week

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Dankook University Hospital, Cheonan, Chungcheongnam-do
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Kyungpook National University Hospital, Daegu, Gyeong Sangbuk-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Yeungnam University Hospital, Daegu, Gyeongsangbuk-do
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hospital, Gwangju, Jeollanam-do
  - Konkuk University Chungju Hospital, Chungju, North Chungcheong